CLINICAL TRIAL: NCT05990036
Title: The Outcome of Sports Vision Training on Collegiate Softball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-1225-EXP
Record Dates: First submitted 2023-06-22; First posted 2023-08-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Athletic Performance
Keywords: Sports; Vision; Training

STUDY DESIGN:
Intervention Model Description: Prospective single cohort with no control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sports vision participants (Experimental): Women softball team participating in a sports vision training program
  Interventions: Other: Sports vision enhancement training curriculum

INTERVENTIONS:
Other: Sports vision enhancement training curriculum — A curriculum of 8 sports vision training procedures applied during women's collegiate softball team training. The training protocol consists of once weekly training sessions, 45 minutes in duration.

SUMMARY:
To investigate the outcomes of sports vision enhancement training on softball players, specifically the visual skills and visual function. This will help to develop and hone best practice methods for future research as well as training protocols for athletes.

DETAILED DESCRIPTION:
After informed consent is given by each participant, they will go through a pre-training evaluation at the Sports Vision Clinic at University Incarnate Word. The evaluation will include a Senaptec Sensory station evaluation of 10 skills, 1) visual acuity 2) contrast sensitivity 3) depth perception 4) near far quickness 5) perception span 6) multiple object tracking 7) reaction time 8) target capture 9) eye hand coordination 10) go/No go. Other skills will be evaluated and re-measured using different types of equipment for better reliability. 11) visual acuity using Rabin Super vision 12) contrast sensitivity using Pelli-Robson and Rabin Super vision 13) accommodative facility 14) reaction time on Dynavision 15) depth perception on the Howard-Dolman, Randot and Automated Vision Tester 16) vergence ranges 17) accommodative amplitude. At the first evaluation each participant will also be asked to complete an entering questionnaire, and at the last evaluation each participate will be asked to complete an exit questionnaire.

The above-mentioned evaluation of 17 items, will be given to each participant pre-training protocol, post-training protocol and once more after a washout period of 5 weeks.

The training protocol will consist of once weekly training sessions 45 minutes in duration. Every participant will receive the same training protocol the only variation will be level of advancement, some athletes will advance at different rates onto more complex levels of each activity. This is to allow continued improvement of the athletes and maintain motivation. Each training session will consist of the following activities 1) Brock string to improve vergence accuracy and depth perception; 2) Senaptec Strobe glasses while performing toss and catch, to improve concentration and visualization; 3) Eye Metrix double eye speed scanning, activities using a number board, aimed at collecting visual information quickly and accurately; 4) Senaptec Synchrony activities to improve anticipation and timing; 5) Senaptec Sensory Station Near Far, focus and concentration activities to improve eye accommodation accuracy; 6) Dynavision activities to improve reaction time, eye-hand coordination, and central-peripheral processing speeds; 7) Sports Vision Trainer Go/No go activities to improve low contrast and go/ no go decision making; 8) Senaptec Sensory Station spatial memory activities to improve memory span and peripheral awareness. Each activity will be performed twice.

ELIGIBILITY:
Inclusion Criteria:

* Member of the University women's softball team
* Pregnancy allowable
* Good academic standing

Exclusion Criteria:

* History of epilepsy
* History of seizures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Target accuracy | Change from baseline at pre-evaluation week 1; to post evaluation at week 12
  An evaluation to compare how many buttons pressed on Dynavision in one minute to the baseline performed at the study onset.
Reaction time | Change from baseline at pre-evaluation week 1; to post evaluation at week 12
  An evaluation to compare average reaction time of buttons pressed on Dynavision in one minute to the baseline performed at the study onset.
Vergence ranges | Change from baseline at pre-evaluation week 1; to post evaluation at week 12
  An evaluation to compare vergences ranges to the baseline performed at the study onset measured by using free space prism ranges distance and near.

SECONDARY OUTCOMES:
Diminished skills; such as Target accuracy, reaction time, vergences ranges. | Change from post evaluation at week 12 compared to final washout evaluation at week 18.
  To see if 5-6 weeks of not training diminishes visual skills trained.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Woideck, DO, Principal Investigator — University of the Incarnate Word
Locations (1):
- University of the Incarnate Word, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zwierko T, Puchalska-Niedbal L, Krzepota J, Markiewicz M, Wozniak J, Lubinski W. The Effects of Sports Vision Training on Binocular Vision Function in Female University Athletes. J Hum Kinet. 2015 Dec 30;49:287-96. doi: 10.1515/hukin-2015-0131. eCollection 2015 Dec 22. PMID 26925183
- [Background] Kutzner BL, Ring M, Michelson G. [Binocular vision training for professional athletes]. Ophthalmologie. 2022 Jul;119(7):721-729. doi: 10.1007/s00347-022-01574-x. Epub 2022 Feb 2. German. PMID 35107596
- [Background] Kirscher DW. Sports vision training procedures. Optom Clin. 1993;3(1):171-82. PMID 8324323
- [Background] Zimmerman AB, Lust KL, Bullimore MA. Visual acuity and contrast sensitivity testing for sports vision. Eye Contact Lens. 2011 May;37(3):153-9. doi: 10.1097/ICL.0b013e31820d12f4. PMID 21378574
- [Background] Formenti D, Duca M, Trecroci A, Ansaldi L, Bonfanti L, Alberti G, Iodice P. Perceptual vision training in non-sport-specific context: effect on performance skills and cognition in young females. Sci Rep. 2019 Dec 10;9(1):18671. doi: 10.1038/s41598-019-55252-1. PMID 31822740
- [Background] Laby DM, Appelbaum LG. Review: Vision and On-field Performance: A Critical Review of Visual Assessment and Training Studies with Athletes. Optom Vis Sci. 2021 Jul 1;98(7):723-731. doi: 10.1097/OPX.0000000000001729. PMID 34328451
- [Background] Hinman SK, Smith KB, Quillen DM, Smith MS. Exercise in Pregnancy: A Clinical Review. Sports Health. 2015 Nov-Dec;7(6):527-31. doi: 10.1177/1941738115599358. Epub 2015 Aug 4. PMID 26502446

DOCUMENTS (3):
  • Study Protocol (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT05990036/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT05990036/SAP_001.pdf
  • Informed Consent Form (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT05990036/ICF_002.pdf